CLINICAL TRIAL: NCT03532503
Title: Second Trimester Pregnancy Termination With Foley Catheter With 30 ml vs 50 ml: Prospective Randomised Study
Brief Title: Second Trimester Pregnancy Termination With Foley Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018.4.18
Record Dates: First submitted 2018-05-09; First posted 2018-05-22 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-05

CONDITIONS: Pregnancy Termination
Keywords: pregnancy termination; second trimester; foley catheter

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foley catheter filled with 30 ml (Active Comparator): The transcervical placement of the foley catheter will be performed and it will be filled with 30 ml saline. A gentle traction will be applied.
  Interventions: Device: Foley catheter
- Foley catheter filled with 50 ml (Active Comparator): The transcervical placement of the foley catheter will be performed and it will be filled with 50 ml saline. A gentle traction will be applied.
  Interventions: Device: Foley catheter

INTERVENTIONS:
Device: Foley catheter — Transcervical foley catheter will be applied

SUMMARY:
One of the methods used to induce second trimester pregnancy termination is the placement of a transcervical Foley catheter. The aim of this randomized controlled study was to assess in pregnant women with an unfavourable cervix, whether there is a difference in efficacy between the two most commonly used insufflation volumes of Foley catheter (30mL and 50mL).

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* second trimester pregnancy ermination

Exclusion Criteria:

* multiple pregnancies

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
induction abortus interval | up to five days
  time to abortus will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided